CLINICAL TRIAL: NCT04358432
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Phase II Study of AK102 in the Treatment of Hypercholesterolemia Patients at Very High or High Risk of Cardiovascular Disease
Brief Title: A Study of PCSK9 Inhibitor AK102 in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: AD Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK102-203
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- AK102 450 mg (Experimental): Participants received AK102 450 mg subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- AK102 300 mg (Experimental): Participants received AK102 300 mg subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- AK102 150 mg (Experimental): Participants received AK102 150 mg subcutaneous injection once every 2 weeks (Q2W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- AK102 75 mg (Experimental): Participants received AK102 75 mg subcutaneous injection once every 2 weeks (Q2W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- Placebo Q4W (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: Placebos; Drug: Statins and/or Ezetimibe
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks
  Interventions: Drug: Placebos; Drug: Statins and/or Ezetimibe

INTERVENTIONS:
Drug: AK102 — Administered by subcutaneous injection
  Arms: AK102 150 mg; AK102 300 mg; AK102 450 mg; AK102 75 mg
Drug: Placebos — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo Q4W
Drug: Statins and/or Ezetimibe — Lipid-lowering therapies

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multicenter study to evaluate the safety and efficacy of AK102 in patients with Hypercholesterolemia Patients at Very High or High Risk of Cardiovascular Disease .

The primary objective of this study is to evaluate the efficacy of AK102 in patients with Hypercholesterolemia Patients at Very High or High Risk of Cardiovascular Disease .

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form (ICF), and be able to comply with the treatment plan, visit, laboratory examination and other requirements specified in the study;
2. Age ≥ 18, male or female;
3. According to the guidelines for the prevention and treatment of dyslipidemia in Chinese adults (revised in 2016), subjects assessed as very high risk or high risk of cardiovascular disease;
4. Subjects received stable and optimal dose of statins for at least 4 weeks before randomization, either in combination with or without ezetimibe;
5. The blood lipid level of the patients with stable 4-week basic lipid-lowering drug treatment met one of the following conditions by the central laboratory test: LDL-C level in very high risk subjects > 1.8 mmol / L (70 mg / dl) or LDL-C level of high-risk subjects > 2.6 mmol / L (100 mg / dl)
6. TG ≤ 4.5 mmol / L (400 mg / dl) measured by central laboratory at screening；

Exclusion Criteria:

1. Has received cholesterol ester transfer protein (CETP) inhibitor within12 months prior to randomization;
2. Has received PCSK9 inhibitors or are known to be allergic to PCSK9 inhibitors or their components;
3. Has received other investigational drugs within 4 weeks or within 5 half lives (whichever was longer) prior to screening.
4. Has previously received biological agent treatment, organ transplantation or gene therapy;
5. Abnormal laboratories prior to the first study drug administration: ALT or AST> 3 × ULN; Creatine kinase > 5 × ULN; eGFR <= 30 ml/min/1.73m2 by Cockcroft Gault method;
6. Uncontrolled hypothyroidism or hyperthyroidism defined as TSH < 1.0 ×LLN or > 1.5 × ULN, respectively;
7. Myocardial infarction, unstable angina pectoris, percutaneous coronary intervention (PCI), coronary bypass grafting (CABG), stroke, severe deep vein thrombosis or pulmonary embolism, or severe arrhythmia occurred within three months prior to randomization ;
8. Grade III or IV according to NYHA assessment;
9. Planned to have heart-related surgery within 3 months after randomization;
10. Type 1 diabetes or poorly controlled type 2 diabetes [HbA1c > 8.5% within 1 month];
11. Subjects with hypertension that could not be controlled by drugs;
12. Known concomitant diseases that may lead to secondary hyperlipidemia, including nephrotic syndrome, cholestatic liver failure, etc;
13. Positive HBsAg or HCV antibody;
14. Known history of primary immunodeficiency virus infection or positive human immunodeficiency virus (HIV) test;
15. History of drug or alcohol abuse prior to screening;
16. Has taken the following drugs within 6 weeks prior to screening: red koji rice > 200 mg/day; niacin > 1000 mg/day; omega-3 fatty acids; steroids or prescription lipid regulating drugs ; cholesterol lowering drugs, health care products, Chinese patent medicines or other food additives other than statins and ezetimibe;
17. Has taken the following drugs within 3 months prior to screening: systemic cyclosporine, systemic steroids, vitamin A derivatives and retinol derivatives for the treatment of skin diseases (such as retinoic acid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 12 | At baseline and week 12

SECONDARY OUTCOMES:
Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) | From baseline through 12 weeks
Percent change from baseline in high-density lipoprotein cholesterol (HDL-C) | From baseline through 12 weeks
Percent change from baseline in non High-density lipoprotein (non-HDL) cholesterol | From baseline through 12 weeks
Percent change from baseline in serum Triglyceride (TG) cholesterol | From baseline through 12 weeks
Percent change from baseline in Apolipoprotein B (Apo B) | From baseline through 12 weeks
Percent change from baseline in Apolipoprotein A-I (ApoA-I) | From baseline through 12 weeks
Percent change from baseline in Lipoprotein(a) [Lp-(a)] | From baseline through 12 weeks
Percent change from baseline in Total Cholesterol(TC) | From baseline through 12 weeks
Incidence of treatment-emergent adverse events | From baseline through 12 weeks
Serum concentrations of AK102 | From baseline through 12 weeks
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline through 12 weeks
  The immunogenicity of AK102 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies.
Change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Principal Investigator — Zhong Shan Hospital Fu Dan University
Locations (2):
- China (2):
  - Zhong Shan Hosipital Fu Dan University, Shanghai
  - Affiliated hospital of Guangdong medical university, Zhanjiang

IPD SHARING:
Plan to Share IPD: No